CLINICAL TRIAL: NCT01600833
Title: To Association of Serum Ferrtin and Homocysteine Levels With Insulin Resistence and Metabolic Syndrome in Women With Polycystic Ovary Syndrome
Brief Title: The Association of Ferrtin and Homocysteine Etc. With RI and MS in Polycystic Ovary Syndrome (PCOS)
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Ming-I Hsu, Taipei Medical University WanFang Hospital, Taipei Medical University WanFang Hospital
Other Study IDs: WFH-TMU-PCOS-201111006
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; Ferritin; Homocysteine; Insulin Resistance; Metabolic Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obese women: BMI>25
- Non obese women: BMI<25

SUMMARY:
The purpose of this study is to study the association of serum ferritin and homocysteine levels with insulin resistance and metabolic syndrome in women with polycystic ovary syndrome The polycystic ovary syndrome (PCOS) is a common endocrine disease, affecting 5-10% of women with reproductive age. Insulin resistance and metabolic disturbance are well-known long-term consequence of women with PCOS. Recent evidence suggests that increased body iron might be involved in the pathogenesis of insulin-resistance disorders, furthermore, hyperhomocysteinemia is associated with an increased risk of atherosclerotic and thromboembolic disorder. The investigators plan to retrospectively review the medical records of female patients who visited the Reproductive Endocrinology Clinic at the Wan Fang Medical Center at Taipei Medical University from Jan 1, 2008, to November 30, 2011.

ELIGIBILITY:
Inclusion Criteria:

* female patients who had been performed with fully PCOS-related survey Who visited the Reproductive Endocrinology Clinic at the Wan Fang Medical Center at Taipei Medical University from Jan 1, 2008, to November 30, 2011.

Exclusion Criteria:

* women who had been diagnosed with disorders of the uterus (e.g., Asherman's Syndrome, Mullerian agenesis), and chromosomal anomalies (e.g., Turner syndrome)
* women who had menopause
* women with inadequate clinical/biochemical records
* women who had had ovarian cysts or ovarian tumors
* women who took hormone, medicine for Diabetes and/or cardiovascular disease.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female patients who had been performed with fully PCOS-related survey Who visited the Reproductive Endocrinology Clinic at the Wan Fang Medical Center at Taipei Medical University from Jan 1, 2008, to November 30, 2011.
Sampling Method: Non-Probability Sample
Enrollment: 539 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Serum ferritin levels in obese and non-obese women. | the patients have PCOS who visited the Reproductive Endocrinology Clinic at the WanFang Medical Center from Jan 1, 2008 to Nov 30, 2011.
  The pathogenesis of increased iron stores correlated with insulin resistance and metabolic syndrome among obese and non-obese premenopausal women was different. The hypertriglyceridemia in women with PCOS might be associated with iron metabolism.

CONTACTS AND LOCATIONS:
Overall Officials: Ming I Hsu, MD, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- WanFang Medical Center at Taipei Medical University, Taipei, Taiwan, Taiwan